CLINICAL TRIAL: NCT02546908
Title: A Multicenter, Prospective, Longitudinal Registry of Patients With Prostate Cancer in Asia
Brief Title: A Registry of Participants With Prostate Cancer in Asia
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR107351; NOPRODPCR4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic Neoplasms; Non-interventional; Observational
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High-risk localized Prostate Cancer (PC): No intervention will be administered in this study. Participants with High-risk localized PC will be enrolled. High-risk localized PC involves clinical T stage greater than or equal to (>=) cT3a and one of the following high risk features: Gleason score 8-10 or prostate specific antigen (PSA) level above 20 nanogram per milliliter (ng/mL).
  Interventions: Other: No Intervention
- Non-metastatic Biochemically Recurrent PC: No intervention will be administered in this study. Participants with Non-metastatic biochemically recurrent PC will be enrolled. A non-metastatic biochemically recurrent PC involves a confirmed PSA value of >0.2 ng/mL following prostatectomy (European Association of Urology (EAU) guidelines), a PSA value of 2 ng/mL or more above the nadir following radiation therapy (American Society for Radiation Oncology (ASTRO) guidelines).
  Interventions: Other: No Intervention
- Metastatic PC: No intervention will be administered in this study. Participants with Metastatic PC will be enrolled.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is an observational study. No study medication is provided will be provided as part of participation. Participants disease status, overall survival (OS), PFS, MFS, SRE-free survival, and time to castration (TTC) will be analyzed according to treatments prescribed while enrolled in the registry. All treatment decisions will be made at the discretion of the investigator or treating physician.

SUMMARY:
The purpose of this study is to document prostate cancer (PC) management including diagnosis, prognosis, treatment, and care in real-world practice.

DETAILED DESCRIPTION:
This is a multicenter (when more than one hospital or medical school team work on a medical research study), prospective (observation of a population for a sufficient number of persons over a sufficient number of years to generate incidence or mortality rates subsequent to the selection of the study group), longitudinal, observational registry (clinical study in which participants may receive diagnostic, therapeutic, or other types of interventions, but the investigator does not assign participants to specific interventions [as in an interventional study])of PC participants. The following 3 participant cohorts will be enrolled: high-risk localized PC, non-metastatic biochemically recurrent PC, and metastatic PC. This is an observational study and treatment decisions and clinical management of participants will follow routine clinical practice. Medical care given to participants will not be influenced by participation in the study. Enrolled participants will be prospectively followed throughout their course of treatment, during which data on PC treatment, clinical progression, and outcomes (including death) will be collected. At the end of registry medical resource utilization (MRU) will also be collected. The maximum observational period will be 5 years. Safety will be monitored throughout the study for participants being treated with JNJ products.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 21 years or older
* Documented diagnosis of PC with either: High-risk localized PC; Non-metastatic, biochemically recurrent PC; Metastatic PC
* Signed participation agreement/Informed Consent Form (ICF) by the patient or a legally acceptable representative
* Agree to be followed-up for PC per routine clinical care

Exclusion Criteria:

* No specific exclusion criteria's were defined

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with High-risk localized prostate cancer (PC), Non-metastatic, biochemically recurrent PC and Metastatic PC will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 3644 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | up to 5 years
  Overall survival is defined as the time from enrollment to date of death due to any cause.
Prostate Cancer (PC)-related Mortality (PM) | up to 5 years
  PC-related mortality is the death due to prostate cancer.
Metastasis-free survival (MFS) | up to 5 years
  MFS is defined as the time from enrollment to the date of the first occurrence of radiographic bone or soft tissue distant metastasis, incidental pathologic finding of distant metastasis, or death from any cause, whichever occurs first.
Progression-free Survival (PFS) | up to 5 years
  Progression-free Survival is the time from enrollment to the occurrence of disease progression or death.
Time to Prostate-specific Antigen (PSA) Progression (TTPP) | up to 5 years
  TTPP is defined as time from enrollment to the date of PSA progression. In participants who has PSA level decreased, PSA progression is defined as 25 percent (%) increase (greater than or equal to [>=] 25%) from nadir (lowest value including baseline) and an increase in the absolute value of at least 2 nanogram per milliliter (ng/mL (>=2ng/mL) and is confirmed by a subsequent measurement at least 3 weeks (>=21 days; PCWG2) after the increase. In participants in whom the PSA level had not decreased, PSA progression is defined as 25% increase (>=25%) from baseline and an increase in the absolute value of at least 2ng/mL (>=2ng/mL) after 12 weeks.
European Quality of Life-5 Dimensions, 5 Levels (EQ-5D-5L) Score | up to 5 years
  The EQ-5D-5L is the new 5-level version of EQ-5D. It describes health-related quality of life (HRQoL) states consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each item of the EQ-5D within these dimensions has 5 response options (no problems, slight problems, moderate problems, severe problems, or extreme problems). Data captured by EQ-5D-5L relates to the patient's status at the time of completion, and takes approximately 5 minutes to complete.
Functional Assessment of Cancer Therapy for Prostate Cancer (FACT-P) Score | up to 5 years
  The FACT-P consists of the FACT-General (FACT-G) and a PC-specific subscale. The FACT-G contains a 27-item questionnaire and is composed of 4 dimensions of HRQoL: physical well-being, social/family well-being, emotional well-being, and functional well-being. The PC-specific subscale is composed of 12 items, which span the dimensions of sexual function, bowel/bladder function, and pain. The FACT-P questionnaire has a 7 day recall, and takes approximately 15 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (31):
- China (8):
  - Beijing
  - Guangzhou
  - Hangzhou
  - Shanghai
  - Shenyang
  - Sichuan
  - Suzhou
  - Wuhan
- India (4):
  - Bangalore
  - Delhi
  - Mumbai
  - New Delhi
- Japan (8):
  - Chiba
  - Hirosaki
  - Ikoma
  - Kobe
  - Koshigaya
  - Matsuyama
  - Ōsaka-sayama
  - Suita
- Malaysia (3):
  - Kuala Lumpur
  - Kuching
  - Pulau Pinang
- Singapore, Singapore
- Seoul, South Korea
- Taiwan (3):
  - Kaohsiung City
  - Tainan
  - Taipei
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Songkhla

REFERENCES:
- [Derived] Ye D, Kanesvaran R, Chiong E, Lojanapiwat B, Pu YS, Rawal SK, Aik OT, Zeng H, Chung BH, Ashani MYN, Ohyama C, Kim CS, Hu Z, Tsai YS, Razack AHA, Singh A, Liu Y, Uemura H. UFO registry: final analysis of baseline data from patients with advanced prostate cancer in Asia. Ther Adv Med Oncol. 2024 Nov 23;16:17588359241293393. doi: 10.1177/17588359241293393. eCollection 2024. PMID 39583953
- [Derived] Uemura H, Ye D, Kanesvaran R, Chiong E, Lojanapiwat B, Pu YS, Rawal SK, Abdul Razack AH, Zeng H, Chung BH, Md Yusoff NA, Ohyama C, Kim CS, Leewansangtong S, Tsai YS, Liu Y, Liu W, van Kooten Losio M, Asinas-Tan M. United in Fight against prOstate cancer (UFO) registry: first results from a large, multi-centre, prospective, longitudinal cohort study of advanced prostate cancer in Asia. BJU Int. 2020 Apr;125(4):541-552. doi: 10.1111/bju.14980. Epub 2020 Jan 30. PMID 31868997
- [Derived] Liu Y, Uemura H, Ye D, Lee JY, Chiong E, Pu YS, Razack AHA, Pripatnanont C, Rawal S, Low GKM, Qiu H, Chow WH, Van Kooten Losio M. Prostate cancer in Asia: design of a patient registry to inform real-world treatments, outcomes, and quality of life. Prostate Int. 2019 Sep;7(3):108-113. doi: 10.1016/j.prnil.2018.12.001. Epub 2018 Dec 24. PMID 31485435